CLINICAL TRIAL: NCT03784014
Title: Molecular Profiling of Advanced Soft-tissue Sarcomas. A Phase III Study
Brief Title: Molecular Profiling of Advanced Soft-tissue Sarcomas
Acronym: MULTISARC
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Collaborators: Commissariat A L'energie Atomique (Other Government); Institut Bergonié (Other); Plateforme labellisée Inca - Institut Bergonié, Bordeaux (Unknown); Plateforme labellisée Inca - Hôpital Européen Georges Pompidou, Paris (Unknown); EUCLID Clinical Trial Platform (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: C16-40; 2024-514873-22-00 (EU CTIS Number); 2017-002851-27 (EudraCT Number)
Record Dates: First submitted 2018-12-19; First posted 2018-12-21 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Soft Tissue Sarcoma
Keywords: advanced disease; metastatic disease; Next generation sequencing exome
MeSH Terms: conditions — Sarcoma; Neoplasm Metastasis | interventions — nilotinib; ceritinib; capmatinib; Lapatinib; trametinib; dabrafenib; olaparib; durvalumab; palbociclib; glasdegib; futibatinib; Base Sequence; High-Throughput Nucleotide Sequencing

STUDY DESIGN:
Intervention Model Description: MULTISARC is a randomized multicenter study assessing whether high throughput molecular analysis (next generation sequencing exome - NGS) is feasible in advanced soft tissue sarcoma participants.
  In parallel, MULTISARC aims to assess efficacy of an innovative treatment strategy guided by high throughput molecular analysis, in participants with advanced soft-tissue sarcomas.
  Randomization 1:1 with 1 participant randomized in experimental Arm NGS (treatment strategy based on NGS) and 1 participant randomized in standard Arm No NGS (treatment strategy not based on NGS).
  At the end of first-line treatment, participant's tumor profile of experimental Arm NGS will be discussed within a multidisciplinary tumor board which aims at discussing the genomic profiles and at providing a therapeutic decision for each participant. Participants for whom a targetable genomic alteration has been identified will be proposed to enter in one of the subsequent phase II single-arm sub-trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm No NGS (No Intervention): Patients will be treated by standard first-line systemic treatment and tumor assessment will be performed every 2 cycles during treatment. Thereafter, disease will be managed as per standard care depending on tumor response observed at the end of the first-line treatment.
  Note that for these participants and under specific conditions, subsequent NGS analyses may be allowed within the scope of the trial
- Arm NGS (Experimental): Patients will be treated by standard first-line systemic treatment and tumor assessment will be performed every 2 cycles during treatment. After tumor assessment at the end of first-line systemic treatment and regardless of tumor response as per RECIST v1.1, participants will be discussed within a multidisciplinary tumor board (molecular tumor board-MTB) which aims at discussing the genomic profiles and at providing a therapeutic decision for each participant.
  Patients for whom a targetable genomic alteration has been highlighted will be proposed to enter in a subsequent single-arm phase II sub-trials. Otherwise, thereafter, disease will be managed as per standard care depending on tumor response observed at the end of the first-line treatment
  Interventions: Other: Next Generation sequencing exome
- Arm NGS - Targeted therapy (Experimental): Targeted therapy from a list of 10 targeted treatment strategies, guided by the genomic analyses: Nilotinib capsule per os 400 mg bd, continuous dosing ; Ceritinib capsule per os 450 mg od, continuous dosing; Capmatinib tablet per os 400 mg bd, continuous dosing; Lapatinib tablet per os 1500 mg od, continuous dosing; Trametinib tablet per os 2 mg od, continuous dosing; association of Trametinib tablet per os 2 mg od and Dabrafenib capsule per os 150 mg bd, continuous dosing; association of Olaparib tablet per os 300 mg bd, continuous dosing and Durvalumab intra-veinous 1500 mg on day 1, Q4W; Palbociclib capsule 125 mg od, 3 weeks on/1 week off; Glasdegib tablet per os 300 mg od, continuous dosing; TAS-120 tablet per os 20 mg od, continuous dosing.
  Interventions: Drug: Nilotinib; Drug: Ceritinib; Drug: Capmatinib; Drug: Lapatinib; Drug: Trametinib; Combination Product: Trametinib and Dabrafenib; Combination Product: Olaparib and Durvalumab; Drug: Palbociclib; Drug: Glasdegib; Drug: TAS-120

INTERVENTIONS:
Drug: Nilotinib — Target: KIT, PDGFRA, CSF1R Nilotinib will be administered orally, 400 mg twice daily on a continuous basis. A treatment cycle consists of 4 weeks. Treatment may continue until disease progression or study discontinuation.
  Other Names: TASIGNA
  Arms: Arm NGS - Targeted therapy
Drug: Ceritinib — Target: ALK, ROS. Ceritinib will be administered orally, 450mg once daily on a continuous basis. A treatment cycle consists of 4 weeks. Treatment may continue until disease progression or study discontinuation.
  Other Names: ZYKADIA
  Arms: Arm NGS - Targeted therapy
Drug: Capmatinib — Target: MET. Capmatinib will be administered orally, 400mg twice daily on a continuous basis. A treatment cycle consists of 4 weeks. Treatment may continue until disease progression or study discontinuation.
  Arms: Arm NGS - Targeted therapy
Drug: Lapatinib — Target: ERBB2, EGFR. Lapatinib will be administered orally, 1500mg once daily on a continuous basis. A treatment cycle consists of 4 weeks. Treatment may continue until disease progression or study discontinuation.
  Other Names: TYVERB
  Arms: Arm NGS - Targeted therapy
Drug: Trametinib — Target: KRAS, NRAS, HRAS, PTPN11, NF1, MAP2K. Trametinib will be administered orally, 2 mg once daily on a continuous basis. A treatment cycle consists of 4 weeks. Treatment may continue until disease progression or study discontinuation.
  Other Names: MEKINIST
  Arms: Arm NGS - Targeted therapy
Combination Product: Trametinib and Dabrafenib — Target: KRAS, NRAS, HRAS, PTPN11, NF1, MAP2K, BRAF. Trametinib will be administered orally, 2mg once daily on a continuous basis. Dabrafenib will be administered orally, 150mg twice daily, on a continuous basis.
  A treatment cycle consists of 4 weeks. Treatment may continue until disease progression or study discontinuation.
  Other Names: MEKINIST and TAFINLAR
  Arms: Arm NGS - Targeted therapy
Combination Product: Olaparib and Durvalumab — Target: PDL1, PARP. Olaparib will be administered orally, 300mg twice daily on a continuous basis. Dabrafenib will be administered intraveinously, 1500mg on day 1 every 4 weeks. A treatment cycle consists of 4 weeks. Treatment may continue until disease progression or study discontinuation.
  Other Names: LYNPARZA; MEDI4736
  Arms: Arm NGS - Targeted therapy
Drug: Palbociclib — Target: CDK4, CDK6. Palbociclib will be administered orally, 125mg once daily, 3 weeks on/1 week off.
  A treatment cycle consists of 4 weeks. Treatment may continue until disease progression or study discontinuation.
  Other Names: IBRANCE; PD-0332991
  Arms: Arm NGS - Targeted therapy
Drug: Glasdegib — Target: SMO. Glasdegib will be administered orally, 300 mg once daily on a continuous basis. A treatment cycle consists of 4 weeks. Treatment may continue until disease progression or study discontinuation.
  Other Names: PF-04449913
  Arms: Arm NGS - Targeted therapy
Drug: TAS-120 — Target: FGFR. TAS-120 will be administered orally, 20 mg once daily on a continuous basis. A treatment cycle consists of 3 weeks. Treatment may continue until disease progression or study discontinuation.
  Arms: Arm NGS - Targeted therapy
Other: Next Generation sequencing exome — Both frozentumor material (archived or newly obtained) and blood sample collection will be used for genetic profiling
  Other Names: RNA Seq; NGS; High throughput sequencing
  Arms: Arm NGS

SUMMARY:
MULTISARC is a randomized multicenter study assessing whether high throughput molecular analysis (next generation sequencing exome - NGS) is feasible in advanced/metastatic soft-tissue sarcoma patients, that is, whether NGS can be conducted for a large proportion of patients, with results available within reasonnable delays.

In parallel, MULTISARC aims to assess efficacy of an innovative treatment strategy guided by high throughput molecular analysis (next generation sequencing exome, RNASeq [NGS]) in patients with Advanced/metastatic soft-tissue sarcomas. At the end of first-line treatment, participant's tumor profile of experimental Arm NGS (treatment strategy based on NGS results) will be discussed within a multidisciplinary tumor board which aims at discussing the genomic profiles and at providing a therapeutic decision for each participant. Participants for whom a targetable genomic alteration has been identified will be proposed to enter in one of the subsequent phase II single-arm sub-trial.

DETAILED DESCRIPTION:
Screening phase: frozen tumor sample (archived or newly obtained) and blood sample will be used for genetic profiling. Patients can be considered as pre-eligible for the randomized phase when all genetic material have been received by the Platform.

Randomization phase: the randomization will allocate the following arms with a ratio 1:1:

* experimental Arm NGS : treatment strategy based on NGS results [exome, RNASeq]
* standard Arm No NGS: treatment strategy not based on NGS (Note that for these participants and under specific conditions, subsequent NGS analyses may be allowed within the scope of the trial)

Single-arm phase II sub-trial: at the end of the first-line treatment and regardless of tumor response as per RECIST v1.1, patients randomized in Arm NGS and for whom a targetable alteration has been identified by the Molecular Tumor Board will be considered as pre-eligible for the targeted sub-study. The mandatory post-chemotherapy wash-out period of 21 days will provide time to achieve all the required tests and examinations.

ELIGIBILITY:
Randomized phase

Inclusion Criteria:

* Age ≥ 18 years,
* Histology: soft-tissue sarcoma confirmed by the RRePS Network, as recommended by the French NCI
* Unresectable locally advanced and/or metastatic STS
* No previous systemic treatment for advanced disease,
* ECOG ≤ 1
* Adequate hematological and metabolic functions: Hemoglobin > 9 g/dL and albumin > 30 g/L
* Measurable disease according to RECIST 1.1. At least one site of disease must be uni-dimensionally > 10 mm,
* Availability of suitable frozen archive tumor material obtained from a metastatic lesion or advanced disease (not previously treated), or at least one lesion that can be biopsied for research purpose,
* Archived FFPE block of specimen tumor sampling obtained anytime during disease development for research purpose,
* Eligible to first-line systemic treatment,
* No prior or concurrent malignant disease diagnosed or treated in the last two years before inclusion. Note that patients with in situ carcinoma of the cervix, or adequately treated basal cell or squamous cell carcinoma of the skin, or adequately treated localized prostate cancer, or other localized cancer under maintenance therapy can be included as long as they don't limit assessment of efficacy of first-line systemic therapy,
* Participant with a social security in compliance with the French law,
* Voluntary signed and dated written informed consent prior to any study specific procedure (ICF1)

Exclusion Criteria:

* Radiological evidence of symptomatic or progressive brain metastases,
* Inability to swallow,
* Major problem with intestinal absorption,
* Previous allogeneic bone marrow transplant,
* Evidence of severe or uncontrolled systemic disease (uncontrolled hypertension, active bleeding diatheses, or active Hepatitis B, C and HIV or active autoimmune disease),
* Any condition which in the Investigator's opinion makes it undesirable for the subject to participate in the trial or which would jeopardize compliance with the protocol,
* Individuals deprived of liberty or placed under guardianship
* Pregnant or breast feeding women,
* Men or women refusing contraception,
* Previous enrolment in the present study,
* Any contraindication to first-line chemotherapy treatment.

Phase II Sub-trials

Inclusion Criteria:

* Participants already enrolled in MULTISARC and randomized/switched in Arm "NGS",
* ECOG performance status < 1,
* Measurable disease according to RECIST v1.1,
* Molecular alteration identified by molecular profiling,
* Participants who have received a first-line systemic treatment at the inclusion,
* Participants must have advanced disease and must not be a candidate for other approved therapeutic regimen known to provide significant clinical benefit based on investigator judgement,
* Participants will have had a minimum of 21 days gap from last chemotherapy or immunotherapy or any other pharmacological therapy and/or radiotherapy prior to the first dose of study treatment,
* Women of childbearing potential must have a negative serum pregnancy test within 3 days of enrolment and serum/urine pregnancy test within 24 hours prior to the administration of the study drug,
* Female with child bearing potential and male participants with partners of child bearing potential must be willing to use two effectives forms of contraception (1 highly effective method and 1 barrier method), from beginning 3 weeks before the first dose of investigational product and until 3 months after discontinuing the study.
* Participant with a social security in compliance with the French law,
* Voluntary signed and dated written informed consent (ICF2) prior to any study specific procedure.

Main exclusion Criteria:

* Previous treatment with the targeted therapy,
* No "targetable" genomic alteration generated during the screening phase either due to the lack of alteration or due to ineligible samples for genomic analysis (MULTISARC),
* Participants with total gastrectomy,
* Major surgery within 30 days prior to entry into the study (excluding placement of vascular access) or minor surgery within 14 days of entry into the study,
* History of hypersensitivity to involved study drug(s) or of its excipients,
* Radiological evidence of symptomatic or progressive brain metastases,
* Participant with oral anticoagulation therapy,
* Inability to swallow,
* Major problem with intestinal absorption,
* Any unresolved toxicity NCI CTCAE Grade ≥2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria. Participants with Grade ≥2 neuropathy will be evaluated on a case-by-case basis after consultation with the Sponsor.
* Previous allogeneic bone marrow transplant,
* Altered hematopoietic or organ function,
* Mean resting corrected QT interval (QTcF)>470msec obtained from 3 consecutive ECGs
* Previous or current maligancies of other histologies within the last 2 years, with the exception of in situ carcinoma of the cervix, and adequately treated basal cell or squamous cell carcinoma of the skin and prostate cancer,
* Evidence of severe or uncontrolled systemic disease (uncontrolled hypertension, active bleeding diatheses), active uncontrolled systemic bacterial, viral, or fungal infection > Grade 2 as per NCI CTCAE v5.0
* Chronic or active hepatitis B or hepatitis C. Testing for hepatitis B surface antigen (HBs Ag) and hepatitis B core antibody (anti HBc) will be performed at screening,
* Human immunodeficiency virus (HIV) positive,
* Any condition which in the Investigator's opinion makes it undesirable for the subject to participate in the trial or which would jeopardize compliance with the protocol,
* Individuals deprived of liberty or placed under guardianship,
* Pregnant or breast feeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 603 (Actual)
Dates: Start 2019-10-19 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2026-01-13 (Estimated)

PRIMARY OUTCOMES:
To assess the feasibility of high throughput molecular analysis (next generation sequencing exome [NGS] | 7 weeks
  Feasibility will be defined as the proportion of participants for whom results from NGS are (i) interpretable and (ii) for whom a validated report of exome sequencing including a clinical recommendation from the molecular tumor board is available within 7 weeks (i.e. within at most 49 calendar days) after reception of blood and tumor samples by one of the molecular platform.

SECONDARY OUTCOMES:
Comparison of the efficacy of the 2 treatment strategies (NGS vs No NGS) in terms of 1-year progression-free survival (PFS) | 1 year
  PFS will be defined as the delay from the date of randomization to the date of progression as per RECIST v1.1 (or death, whichever occurs first)
Comparison of the efficacy of the 2 treatment strategies (NGS vs No NGS) in terms of 2-year progression-free survival (PFS) | 2 years
  PFS will be defined as the delay from the date of randomization to the date of progression as per RECIST v1.1 (or death, whichever occurs first)
Comparison of the efficacy of the 2 treatment strategies (NGS vs No NGS) in terms of 1-year overall survival (OS) | 1 year
  OS will be defined as the delay from the date of randomization to the date of death (whatever the cause)
Comparison of the efficacy of the 2 treatment strategies (NGS vs No NGS) in terms of 2-year overall survival (OS) | 2 years
  OS will be defined as the delay from the date of randomization to the date of death (whatever the cause)
Assessment of the feasibility of high throughput molecular analysis in terms of delay to obtain a clinical recommendation from the molecular tumor board for patients randomized in arm NGS with interpretable NGS | an average of 7 weeks
  Delay from the date of signature of the informed consent to the date of the molecular tumor board
Assessment of the proportion of patients with Advanced STS presenting at least one targetable genomic alteration | An average of 7 weeks
  A participant will be considered as "presenting at least one targetable genomic alteration", if the MTB considers that at least one genetic alteration identified can be matched with one of the drugs available through the MULTISARC study
Assessment of the efficacy of first-line systemic treatment in terms of 1-year progression-free survival | 1 year
  PFS will be defined as the delay from the date of onset of first-line treatment to the date of progression as per RECIST v1.1 (or death, whichever occurs first)
Assessment of the efficacy of first-line systemic treatment in terms of 2-year progression-free survival | 2 years
  PFS will be defined as the delay from the date of onset of first-line treatment to the date of progression as per RECIST v1.1 (or death, whichever occurs first)
Assessment of the efficacy of first-line systemic treatment in terms of 1-year overall survival | 1 year
  OS will be defined as the delay from the date of onset of first-line treatment to the date of death (whatever the cause).
Assessment of the efficacy of first-line systemic treatment in terms of 2-year overall survival | 2 years
  OS will be defined as the delay from the date of onset of first-line treatment to the date of death (whatever the cause).
Assessment of the efficacy of first-line systemic treatment in terms of best overall response under first-line treatment | Throughout the treatment period, an average of 18 weeks
  Best response is recorded from the date of onset of first-line treatment until the end of first-line treatment taking into account any requirement for confirmation as per RECIST v1.1 criteria
Assessment of the efficacy of first-line systemic treatment in terms of 6-month objective response | 6 months
  Objective response is defined as complete or partial response (CR, PR) as per RECIST v1.1 under first-line treatment
Assessment of the efficacy of first-line systemic treatment in terms of 6-month non progression | 6 months
  Non progression is defined as complete or partial response (CR, PR) or stable disease (SD) under first-line treatment as defined as per RECIST v1.1
Assessment of the efficacy of each targeted treatment in terms of 6-month non progression | 6 months
  Non progression is defined as complete or partial response (CR, PR) or stable disease (SD) under targeted treatment as defined as per RECIST v1.1
Assessment of the efficacy of each targeted treatment in terms of 1-year progression-free survival | 1 year
  PFS will be defined as the delay from the date of targeted treatment initiation to the date of progression as per RECIST v1.1 or death, whichever occurs first
Assessment of the efficacy of each targeted treatment in terms of 1-year overall survival | 1 year
  OS is defined as the delay from the date of targeted treatment initiation to the date of death (whatever the cause)
Assessment of the efficacy of each targeted treatment in terms of best overall response under treatment | Throughout the treatment period, an average of 6 months
  Best response (partial or complete, as per RECIST v1.1) recorded from date of targeted treatment initiation taking into account any requirement for confirmation as per RECIST v1.1 criteria
Assessment of the efficacy of each targeted treatment in terms of objective response under treatment | Throughout the treatment period, an average of 6 months
  Complete response or partial response under targeted treatment as defined as per RECIST evaluation criteria v1.1
Assessment of the efficacy of each targeted treatment in terms of change in tumor size (CTS) | Throughout the treatment period, an average of 6 months
  CTS is defined as the difference (in percentage) in tumor size burden from the date of targeted treatment initiation (baseline) to the tumor assessment
Assessment of the safety profile of each targeted treatment using the CTCAE v5 | Throughout the treatment period, an average of 6 months
  Safety will be assessed as per CTCAE v5
Impact of the results of immunosequencing during first-line treatment | At cycle 2 day 1 of targeted treatment
  Correlation of TCR-sequencing data with objective response (OR), OR), progression-free survival (PFS) and overall survival (OS).
  Evaluation of the association between immune profiles derived from ancillary analyses (VISIUM HD, multiplex IF, SomaScan proteomics) and treatment response, within an integrated immunosequencing framework.
To estimate the cost-effectiveness of the strategy usdin NGS as compared to the strategy without NGS | Trhoughout the study period, an average of 2 years
  The outcome will be the incremental cost-utility ratio or the incremental cost per incremental Quality Adjusted Life Year (QALY)
To assess the feasibility of NGS in participants who have switched treatment arm for NGS arm in terms of proportion of participants with interpretable NGS results | an average of 7 weeks
  Proportion of participants with interpretable NGS results
To assess the feasibility of NGS in participants who have switched treatment arm for NGS arm in terms of delays | an average of 7 weeks
  Delay from the date of treatment failure (progression, investigator decision, end of last treatment line) to the date of the molecular tumor board
To assess the feasibility of NGS in participants who have switched treatment arm for NGS arm in terms of proportion of participants with interpretable NGS results | an average of 7 weeks
  Proportion of participants presenting at least one targetable genomic alteration

CONTACTS AND LOCATIONS:
Overall Officials: Antoine Italiano, Principal Investigator — Institut Bergonié
Locations (17):
- France (17):
  - Institut Bergonie, Bordeaux
  - Centre Georges François Leclerc, Dijon
  - Centre Oscar Lambret, Lille
  - Centre Léon Bérard, Lyon
  - Institut Paoli Calmettes, Marseille
  - Institut de Cancérologie de Montpellier, Montpellier
  - Centre Antoine Lacassagne, Nice
  - Hôpital Cochin, Paris
  - Hôpital Pitié Salpétrière, Paris
  - Institut Curie, Paris
  - CHU Poitiers, Poitiers
  - Centre Eugène Marquis, Rennes
  - Centre Henri Becquerel, Rouen
  - Institut de Cancérologie de l'Ouest - Site René Gauducheau, Saint-Herblain
  - ICANS - Institut de Cancérologie Strasbourg, Strasbourg
  - IUCT Oncopôle, Toulouse
  - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: Yes
Data from the MULTISARC study will be integrated into the Data Collector and Analyzer (CAD) provided for the Plan for Personalized Genomic Medicine 2025, where they will be stored for use in diagnostic and prognostic decision support, the development of therapeutic strategies, and health-related research, studies and evaluations.
  Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of scientific and ethic commitee of the CAD.

REFERENCES:
- [Background] Italiano A. Is There Value in Molecular Profiling of Soft-Tissue Sarcoma? Curr Treat Options Oncol. 2018 Dec 7;19(12):78. doi: 10.1007/s11864-018-0589-y. PMID 30523434
- [Result] FGM 2025 Workflow Study Group (Alliance nationale des Sciences de la Vie et de la Sante); Auzanneau C, Bacq D, Bellera C, Blons H, Boland A, Boucheix M, Bourdon A, Chollet E, Chomienne C, Deleuze JF, Delmas C, Dinart D, Esperou H, Geillon F, Geneste D, Italiano A, Jean D, Khalifa E, Laizet Y, Laurent-Puig P, Lethimonnier F, Levy-Marchal C, Lucchesi C, Malle C, Mancini P, Mathoulin-Pelissier S, Meyer V, Marie-Ange P, Perkins G, Sellan-Albert S, Soubeyran I, Wallet C. Feasibility of high-throughput sequencing in clinical routine cancer care: lessons from the cancer pilot project of the France Genomic Medicine 2025 plan. ESMO Open. 2020 Jul;5(4):e000744. doi: 10.1136/esmoopen-2020-000744. PMID 32713836
- [Result] Italiano A, Dinart D, Soubeyran I, Bellera C, Esperou H, Delmas C, Mercier N, Albert S, Poignie L, Boland A, Bourdon A, Geneste D, Cavaille Q, Laizet Y, Khalifa E, Auzanneau C, Squiban B, Truffaux N, Olaso R, Gerber Z, Wallet C, Benard A, Blay JY, Laurent-Puig P, Deleuze JF, Lucchesi C, Mathoulin-Pelissier S; MULTISARC study group. Molecular profiling of advanced soft-tissue sarcomas: the MULTISARC randomized trial. BMC Cancer. 2021 Nov 5;21(1):1180. doi: 10.1186/s12885-021-08878-2. PMID 34740331